CLINICAL TRIAL: NCT04896697
Title: A First-in-Human, Multicenter, Phase 1/2, Open-Label Study of Vilastobart (XTX101) Monotherapy and Vilastobart (XTX101) and Atezolizumab Combination Therapy in Patients With Advanced Solid Tumors
Brief Title: Vilastobart (XTX101) Monotherapy and Vilastobart and Atezolizumab Combination Therapy in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xilio Development, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XTX101-01/02-001
Record Dates: First submitted 2021-05-06; First posted 2021-05-21 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1A - vilastobart (XTX101) Monotherapy Dose Escalation (Experimental): Part 1A Dose Escalation of vilastobart (XTX101) administered in ascending doses to patients with advanced or metastatic solid tumors to find the recommended phase 2 dose (RP2D).
  Interventions: Drug: vilastobart (XTX101)
- Part 1B - Pharmacodynamic (PD) Dose Expansion (Experimental): Part 1B vilastobart (XTX101) at the RP2D will be administered to further examine vilastobart (XTX101) as monotherapy in patients with select advanced solid tumors.
  Interventions: Drug: vilastobart (XTX101)
- Part 1C - vilastobart (XTX101) Dose Escalation and Dose Expansion in Combination with Atezolizumab (Experimental): Part 1C will receive a labeled dose of atezolizumab in combination with vilastobart (XTX101).
  Interventions: Drug: Atezolizumab; Drug: vilastobart (XTX101)
- Phase 2 - vilastobart (XTX101) Dose Expansion in Combination with Atezolizumab (Experimental): Phase 2 will receive a labeled dose of atezolizumab in combination with vilastobart (XTX101) at the RP2D(s) in patients with MSS CRC.
  Interventions: Drug: Atezolizumab; Drug: vilastobart (XTX101)

INTERVENTIONS:
Drug: vilastobart (XTX101) — vilastobart (XTX101) monotherapy
  Arms: Part 1A - vilastobart (XTX101) Monotherapy Dose Escalation; Part 1B - Pharmacodynamic (PD) Dose Expansion
Drug: Atezolizumab — 1200 mg administered every 3 weeks in combination with vilastobart (XTX101)
  Arms: Part 1C - vilastobart (XTX101) Dose Escalation and Dose Expansion in Combination with Atezolizumab; Phase 2 - vilastobart (XTX101) Dose Expansion in Combination with Atezolizumab
Drug: vilastobart (XTX101) — In combination with Atezolizumab
  Arms: Part 1C - vilastobart (XTX101) Dose Escalation and Dose Expansion in Combination with Atezolizumab; Phase 2 - vilastobart (XTX101) Dose Expansion in Combination with Atezolizumab

SUMMARY:
This is a first-in-human, Phase 1/2, multicenter, open-label study designed to evaluate the safety and tolerability of vilastobart (XTX101) as monotherapy and vilastobart (XTX101) and atezolizumab combination therapy in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1/2, multicenter, open-label study designed to evaluate the safety and tolerability of vilastobart (XTX101), a tumor-selective anti-CTLA-4 antibody, as monotherapy and vilastobart (XTX101) and atezolizumab combination therapy in patients with advanced solid tumors.

Part 1A will examine vilastobart (XTX101) monotherapy in an accelerated and standard 3+3 dose escalation design. Based on the results of Part 1A, patients with select advanced solid tumors will be enrolled in Part 1B, which will evaluate vilastobart (XTX101) monotherapy in relation to specific PD biomarkers.

Part 1C will examine vilastobart (XTX101) in combination with atezolizumab in a standard 3+3 dose escalation/dose de-escalation design. Part 1C may include a dose expansion cohort to further evaluate the safety, PK, and PD of dose levels that were previously cleared.

Phase 2 will examine vilastobart (XTX101) in combination with atezolizumab in patients with metastatic microsatellite stable colorectal cancer (MSS CRC) at the RP2D(s) defined in Part 1C.

ELIGIBILITY:
Inclusion Criteria:

Disease Criteria -

* Part 1A and 1C: Any histologically or cytologically confirmed solid tumor malignancy that is locally advanced or metastatic and has failed standard therapy, or standard therapy is not curative or available;
* Part 1B:

  * Any histologically or cytologically confirmed solid tumor malignancy for which anti-PD-1 or anti-PD-L1 treatment is approved and has progressed on or after prior anti-PD-1 or anti-PD-L1 therapy.
  * Patients with metastatic castrate-resistant prostate cancer if they have progressed on at least 2 lines of systemic therapy
  * Patients with extensive stage small cell lung cancer (SCLC) after at least 1 line of prior therapy
  * Patients with microsatellite stable colorectal cancer after at least 2 lines of prior therapy
* Phase 2: Patients with histologically confirmed metastatic MSS CRC are eligible to enroll in Phase 2 as follows:

  * Patients must have had at least 1 prior chemotherapy regimen for metastatic CRC including all of the following agents: a fluoropyrimidine, irinotecan, oxaliplatin, bevacizumab or biosimilars, an anti epidermal growth factor receptor antibody (cetuximab or panitumumab), and v-raf murine sarcoma viral oncogene homolog B1 inhibitor/BRAF (encorafenib), if applicable
  * Patients with MSI-H/dMMR are excluded
* ECOG performance status of 0 or 1
* Adequate organ function
* Part 1B, Part 1C, and Phase 2 only: measurable disease per iRECIST

Exclusion Criteria:

* Received prior treatment with anti-CTLA-4 therapy
* Received prior immune-checkpoint therapy and experienced Grade 3 or greater toxicity lasting greater than 6 weeks
* Received prior approved systemic anticancer therapy within 4 weeks prior to study treatment
* Received prior radiotherapy within 2 weeks prior to study treatment
* Phase 2 only: Received prior anti-PD-1/L1 therapy or any investigational checkpoint inhibitory therapy
* Has a diagnosis of immunodeficiency
* Has known malignancy (other than disease under study) that is progressing or has required active treatment within the past 3 years
* Has an active autoimmune disease that has required systemic treatment in past 2 years, including the use of disease modifying agents, corticosteroids or immunosuppressive drugs
* Has an active infection requiring systemic intravenous therapy within 4 weeks prior to study treatment, or oral therapy within 2 weeks prior to study treatment
* Has a history of severe hypersensitivity reaction (≥ Grade 3) to any study intervention and/or any of its excipients
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Phase 2 only: symptomatic bowel obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) in Part 1A | Cycle 1 Day 1 up to just prior to the second dose of study drug at Cycle 2 day 1 (approximately 3 weeks)
Incidence of Dose Limiting Toxicities (DLTs) in Part 1C | Cycle 1 Day 1 up to Cycle 3 Day 1 (approximately 6 weeks)
Incidence of treatment-emergent adverse events in Part 1 | Up to 24 months
Incidence of changes in clinical laboratory abnormalities in Part 1 | Up to 24 months
Investigator-assessed objective response rate (ORR) per iRECIST in Phase 2 | Up to 24 months

SECONDARY OUTCOMES:
Investigator-assessed objective response rate (ORR) per iRECIST in Part 1 | Up to 24 months
Antidrug antibody (ADA) occurrence and titer in serum in Part 1 | Up to 24 months
Plasma concentrations of vilastobart (XTX101) (total and intact) in Part 1 and Phase 2 | Up to 24 months
Maximum observed plasma concentration (Cmax) in Part 1 and Phase 2 | Up to 24 months
Time of maximum observed concentration (Tmax) in Part 1 and Phase 2 | Up to 24 months
Trough concentrations (Ctrough) in Part 1 and Phase 2 | Up to 24 months
Area under the curve (AUC) in Part 1 and Phase 2 | Up to 24 months
Half-life (T1/2) in Part 1 and Phase 2 | Up to 24 months
Systemic clearance (CL) in Part 1 and Phase 2 | Up to 24 months
Volume of distribution (Vd) in Part 1 and Phase 2 | Up to 24 months
Investigator-assessed ORR per RECIST in Phase 2 | Up to 24 months
Duration of response per iRECIST in Phase 2 | Up to 24 months
  The time from first documented confirmed response to first documented disease progression
Disease control rate in Phase 2 | Up to 24 months
  The percent of patients who achieve complete response per iRECIST (iCR), partial response per iRECIST (iPR), or stable disease per iRECIST (iSD)
Progression-free survival per iRECIST in Phase 2 | Up to 24 months
  The time from first dose to first documented disease progression or death
Overall survival in Phase 2 | Up to 24 months
  The time from first dose to death due to any cause
Incidence of treatment-emergent AEs in Phase 2 | Up to 24 months
Incidence of changes in clinical laboratory abnormalities in Phase 2 | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - California Cancer Associates for Research and Excellence, cCARE, Encinitas, California
  - City of Hope-Lennar, Irvine, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - California Cancer Associates for Research and Excellence, cCARE, San Marcos, California
  - UCLA Hematology/Oncology- Santa Monica, Santa Monica, California
  - City of Hope-Upland, Upland, California
  - Mayo Clinic Hospital, Jacksonville, Florida
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Orlando, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic Hospital, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - University of Pittsburgh Medical Center- Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Next Oncology, Austin, Texas
  - Mary Crowley Cancer Research, Dallas, Texas
  - Tranquil Clinical Research, Webster, Texas
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jenkins KA, Park M, Pederzoli-Ribeil M, Eskiocak U, Johnson P, Guzman W, McLaughlin M, Moore-Lai D, O'Toole C, Liu Z, Nicholson B, Flesch V, Qiu H, Clackson T, O'Hagan RC, Rodeck U, Karow M, O'Neil J, Williams JC. XTX101, a tumor-activated, Fc-enhanced anti-CTLA-4 monoclonal antibody, demonstrates tumor-growth inhibition and tumor-selective pharmacodynamics in mouse models of cancer. J Immunother Cancer. 2023 Dec 12;11(12):e007785. doi: 10.1136/jitc-2023-007785. PMID 38164757